CLINICAL TRIAL: NCT07189507
Title: Evaluation of the 26 °C Indoor Temperature Upper Limit Considering Clothing Insulation and Daily Activity in Older Adults
Brief Title: Suitability of the 26 °C Indoor Temperature Upper Limit for Older Adults: Impacts of Clothing and Daily Activity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Glen P. Kenny, Full Professor, University Research Chair, University of Ottawa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HEPRU-2025-09-A
Record Dates: First submitted 2025-09-16; First posted 2025-09-24 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Heat Stress; Physiological Stress
Keywords: Indoor overheating; Indoor temperatures; Heat wave; Thermoregulation; Heat strain; Heat vulnerability; Hyperthermia; Elderly; Thermal comfort; Clothing; Activity
MeSH Terms: conditions — Heat Stress Disorders; Hyperthermia; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exposure to indoor temperature upper limit without physical activity and added clothing. (Experimental): Participants, dressed in light clothing (t-shirt, shorts and socks), perform seated rest while exposed daylong (8 hours) to an indoor temperature maintained at 26°C and 45% relative humidity (humidex equivalent of 29).
  Interventions: Other: Simulated indoor temperature upper limit
- Exposure to indoor temperature upper limit with physical activity. (Experimental): Participants, dressed in light clothing (t-shirt, shorts and socks), perform light exercise (i.e., stepping, representing activities of daily living, 4-4.5 METS) every hour (except during lunch hour period) while exposed daylong (8 hours) to an indoor temperature maintained at 26°C and 45% relative humidity (humidex equivalent of 29).
  Interventions: Other: Simulated indoor temperature upper limit
- Exposure to indoor temperature upper limit with added clothing. (Experimental): Participants, dressed in light clothing (t-shirt, shorts and socks) and an added clothing layer (sweatshirt and sweatpants), perform seated rest while exposed daylong (8 hours) to an indoor temperature maintained at 26°C and 45% relative humidity (humidex equivalent of 29).
  Interventions: Other: Simulated indoor temperature upper limit
- Exposure to indoor temperature upper limit with physical activity and added clothing. (Experimental): Participants, dressed in light clothing (t-shirt, shorts and socks) and an added clothing layer (sweat shirt and sweat pants), perform light exercise (i.e., stepping, representing activities of daily living, 4-4.5 METS) every hour (except during lunch hour period) while exposed daylong (8 hours) to an indoor temperature maintained at 26°C and 45% relative humidity (humidex equivalent of 29).
  Interventions: Other: Simulated indoor temperature upper limit

INTERVENTIONS:
Other: Simulated indoor temperature upper limit — Older adults exposed to an 8-hour simulated exposure.

SUMMARY:
While an upper limit of 26°C has been shown to be protective for heat-vulnerable older occupants (DOI: 10.1289/EHP11651), this recommendation did not consider the added heat burden associated with increases in internal heat production accompanying activities of daily living or the restriction to heat loss caused by clothing insulation. To safeguard the health of older adults, health agencies worldwide recommend the remain in cool space indoors, avoid strenuous activity, wear lightweight clothing, and drink cool water regularly throughout the day. However, older adults do not sense heat as well as their younger counterparts. Consequently, they may not take appropriate countermeasures to mitigate physiological strain from indoor overheating. This may include overdressing despite high indoor temperatures. In other cases, individuals may wear insulated clothing in hot weather to observe cultural or religious modesty requirements, which serve as expressions of faith and identity rather than a tool for thermoregulation. Further, individuals may be unaware of the consequences of increases in physical activity on heat gain and may therefore not adjust their normal day-to-day activity levels to prevent potentially dangerous rises in body temperature. Consequently, this may necessitate a lowering of recommended upper indoor temperature limit during hot weather.

To address these important considerations, on separate occasions the investigators will assess the change in body temperature and cardiovascular strain in older adults (65-85 years) exposed for 8 hours to the recommended indoor temperature upper limit of 26°C and 45% relative humidity equivalent humidex of 29 (considered comfortable) while they A) perform seated rest dressed in light clothing (t-shirt, shorts and socks), B) perform light exercise (stepping exercise to simulate activities of daily living, 4-4.5 METS) every hour (except during lunch hour period) dressed in light clothing, C) perform light exercise (4-4.5 METS) every hour (except during lunch hour period) dressed in light clothing (t-shirt, shorts and socks) and an added clothing layer (sweatshirt and sweatpants) and D) perform seated rest dressed in light clothing (t-shirt, shorts and socks) and an added clothing layer (sweatshirt and sweatpants). With this experimental design, investigators will assess the effects of added clothing insulation and light activity, representative in activities of daily living on physiological strain and identify whether refinements in the recommended 26°C indoor temperature limit may be required.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking.
* English or French speaking.
* Ability to provide informed consent.
* with or without a) chronic hypertension (elevated resting blood pressure; as defined by Heart and Stroke Canada and Hypertension Canada), b) type 2 diabetes as defined by Diabetes Canada, with at least 5 years having elapsed since time of diagnosis

Exclusion Criteria:

* Episode(s) of severe hypoglycemia (requiring the assistance of another person) within the previous year, or inability to sense hypoglycemia (hypoglycemia unawareness).
* Serious complications related to your diabetes (gastroparesis, renal disease, uncontrolled hypertension, severe autonomic neuropathy).
* Uncontrolled hypertension - BP >150 mmHg systolic or >95 mmHg diastolic in a sitting position.
* Restrictions in physical activity due to disease (e.g. intermittent claudication, renal impairment, active proliferative retinopathy, unstable cardiac or pulmonary disease, disabling stroke, severe arthritis, etc.).
* Use of or changes in medication judged by the patient or investigators to make participation in this study inadvisable.
* Cardiac abnormalities identified during screening

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Core temperature (Peak) during daylong exposure to indoor temperature limit. | End of 8 hour daylong exposure
  Peak rectal temperature (15 min average) during exposure. Rectal temperature is measured continuously throughout the 8 hour exposure to the simulated indoor temperature upper limit.
Core temperature (AUC) during daylong exposure to indoor temperature limit. | End of 8 hour daylong exposure
  Areas under the curve (AUC) of rectal temperature during the 8 hour exposure to the simulate indoor temperature upper limit.
Core temperature end of daylong exposure to indoor temperature limit. | End of 8 hour daylong exposure
  Rectal temperature measured at hour 8 of exposure to indoor temperature limit (15-min average).
Mean skin temperature (Peak) during daylong exposure to indoor temperature limit. | End of 8 hour daylong exposure
  Peak mean skin temperature (15 min average) during exposure. Mean skin temperature as calculated from skin temperature measured across 7 body regions is measured continuously throughout the 8 hour exposure to the simulated indoor temperature upper limit.
Mean skin temperature (AUC) during daylong exposure to indoor temperature limit. | End of 8 hour daylong exposure
  Areas under the curve (AUC) of mean skin temperature as calculated over 7 body regions during the 8 hour exposure to the simulate indoor temperature upper limit.
Mean skin temperature end of daylong exposure to indoor temperature limit. | End of 8 hour daylong exposure
  Mean skin temperature measured over 7 body regions at hour 8 of exposure to indoor temperature limit (15-min average).
Heat rate (Peak) during daylong exposure to indoor temperature limit. | End of 8 hour daylong exposure
  Peak heart rate (15 min average) during exposure. Heart rate is measured continuously throughout the 8 hour exposure to the simulated indoor temperature upper limit.
Heart rate (AUC) during daylong exposure to indoor temperature limit. | End of 8 hour daylong exposure
  Areas under the curve (AUC) of heart rate during the 8 hour exposure to the simulate indoor temperature upper limit.
Heart rate end of daylong exposure to indoor temperature limit. | End of 8 hour daylong exposure
  Heart rate measured at hour 8 of exposure to indoor temperature limit (15-min average).
Heart rate variability: RMSSD during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Root mean squared standard deviation of normal-to-normal R-wave to R-wave intervals (RMSSD) measured during 5 minutes of paced breathing (15 breaths/min) with participants in the supine position. RMSSD will be evaluated twice, during two paced breathing periods (separated by 4 min of supine rest).
Heart rate variability: SDNN during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Standard deviation of normal-to-normal R-wave to R-wave intervals (SDNN) measured during 5 minutes of paced breathing (15 breaths/min) with participants in the supine position. SDNN will be evaluated twice, during two paced breathing periods (separated by 4 min of supine rest).
Cardiac response to standing from supine (30:15 ratio) during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Cardiac response to standing evaluated as the ratio between the highest R-wave to R-wave interval (lowest heart rate) measured at the 30th heart beat after standing from supine (+/- 5 beats) and the lowest R-wave to R-wave interval (highest heart rate) measured at the 15th heart beat after standing (+/- 5 beats). Cardiac response to standing will be evaluated twice, during two lying-to-standing tests (separated by 10 min of supine rest).
Systolic response to standing from supine during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Systolic blood pressure response to standing evaluated as the difference in blood pressure measured between the standing and supine. Standing systolic blood pressure will be taken as the lowest value of those measured after 60 and 120 seconds of standing. Systolic response to standing will be evaluated twice, during two lying-to-standing tests (separated by 10 min of supine rest).
Systolic blood pressure during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Systolic blood pressure measured in triplicate via automated oscillometry (~60 seconds between measures).
Diastolic blood pressure during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Diastolic blood pressure measured in triplicate via automated oscillometry (~60 seconds between measures).
Rate pressure product during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Rate pressure product, an index of myocardial work and strain, calculated as systolic blood pressure x heart rate.
Reaction time during daylong exposure to indoor temperature limit (cognitive function). | At the start (hour 0) and end of 8 hour daylong exposure
  Participants will be provided with a tablet device with the Sway Medical testing platform for the assessment of reaction time. Participants will be asked to initiate a movement of the device in response to a visual cue.
Impulse control during daylong exposure to indoor temperature limit (cognitive function). | At the start (hour 0) and end of 8 hour daylong exposure
  Participants will be provided with a tablet device with the Sway Medical testing platform for the assessment of impulse control. Participants will be asked to respond to both "go" and "no-go" visual cues. In response to the "go" cue, participants will initiate a movement of the device.
CDC 4-Stage Balance Test during daylong exposure to indoor temperature limit (postural stability). | At the start (hour 0) and end of 8 hour daylong exposure
  To assess postural stability, participants hold a tablet to their chest, then auditory cues guide participants through four consecutive stances, feet side by side, instep of one foot touching the big toe of the other foot, tandem stand with one foot in front of the other, heel touching toe, and stand on one foot. The balance assessment will be evaluated based on movement detected by an accelerometer integrated into the hardware of the tablet device (Sway Medical Inc).
BTrackS Balance Assessment during daylong exposure to indoor temperature limit (postural stability). | At the start (hour 0) and end of 8 hour daylong exposure
  To assess postural stability, participants will be asked to stand on a BTracks force plate with their feet spread out to shoulder width while looking straight ahead. The assessment will comprise of one trial lasting 120 seconds in length. Center of pressure (COP) vector data along vertical (y) and horizontal (x) axes will be summed for the total path excursion length (cm) during each trial.
Fluid consumption during daylong exposure to indoor temperature limit. | At end of 8 hour daylong exposure
  Average hourly fluid consumption calculated by weighing participant water intake at the start and end of each hour of exposure (normalized to the exposure duration).
Fluid loss during daylong exposure to indoor temperature limit. | At end of 8 hour daylong exposure
  Fluid loss calculated as the change in body mass during each exposure presented as a percentage of baseline body mass (corrected for food consumption).
Change in plasma volume during daylong exposure to indoor temperature limit. | At end of 8 hour daylong exposure.
  Change in plasma volume from baseline values calculated from duplicate measurements of hemoglobin and hematocrit at the start and end of each exposure using the technique by Dill and Costill.
Thermal comfort scale during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Thermal comfort assessed via a visual analog scale ("How comfortable does your body temperature feel?") ranging from "very uncomfortable" to "comfortable".
Thirst sensation scale during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Thirst sensation assessed via a visual analog scale ranging from "very, very thirsty" to "not thirsty at all".
Arousal scale during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Felt arousal scale assessed via a visual analog scale ("How worked up are you?") ranging from "high arousal" to "low arousal".
Thermal sensation scale during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Thermal sensation assessed via a visual analog scale ("How hot do you feel?") ranging from "extremely hot" to "neutral"(midpoint: hot)
Thermal sensation 2 scale during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Thermal sensation assessed via a visual analog scale ("How do you feel?") ranging from "hot" to "cold"(midpoint: neutral)
Orthostatic intolerance symptoms assessment during daylong exposure to indoor temperature limit. | At end of 8 hour daylong exposure.
  Cumulative sum of scores on 6 questions asking participant to rank symptoms associated with orthostatic intolerance during the lying to standing tests. All symptoms scored on a scale from 0 (none) to 10 (worst possible) and include feelings of: (1) "dizziness, lightheadedness, feeling faint, or feeling like you might black out"; (2) "Problems with vision (blurring, seeing spots, tunnel vision, etc.)"; (3) "Weakness"; (4) "Fatigue"; (5) "Trouble concentrating"; and (6) "Head and neck discomfort".
Feel good scale during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Feel good assessed via a visual analog scale ("How good do you feel?") ranging from "very good" to "very bad"(midpoint: neutral)
Perceived exertion scale during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Perceived exertional assessed via a visual analog scale ("How hard are you working?") ranging from "no exertional at all" to "maximal exertion"
Hydration status during daylong exposure to indoor overheating | At the start (hour 0) and end of 8 hour daylong exposure
  Hydration status measured via assessing the urine specific gravity of a urine sample.
Activity levels during daylong exposure to indoor overheating | End of 8 hour daylong exposure
  Activity levels assessed via a wearable monitor (Actical) containing an accelerometer worn on the wrist and hip.

SECONDARY OUTCOMES:
Profiles of Mood States (POMS) during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Potential changes in mood (7 subscales of mood: tension, anger, depression, fatigue, confusion, vigor and esteem related affect). The POMS-40 is a validated, self-administered questionnaire that examines seven distinct aspects of mood state across two positive subscales (Esteem-Related Affect, and Vigor) and five negative subscales (Fatigue, Tension, Confusion, Anger, and Depression), which are described across 40 distinct adjectives. For each individual item, participants were asked to describe "how you feel right now" by responding using a 5-point Likert scale (0 = "Not at all", 1 = "A little", 2 = "Moderately", 3 = "Quite a lot", or 4 = "Extremely"). The values of items associated with a specific subscale (e.g., Fatigue) were summed to calculate its score.
Environmental Symptoms Questionnaire (ESQ) during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 8 hour daylong exposure
  Self-reported environmental reactions and medical symptomatology associated with prolonged heat exposure. The ESQ-IV is a validated 68-item, self-administered questionnaire that has been used successfully in identifying symptomatology during exposure to a wide variety of environmental conditions, including heat exposure [24, 25].
  Participants are asked to assess and described "how you have been feeling today" by responding to each item using a 6-point Likert scale (0 = "Not at all", 1 = "Slight", 2 = "Somewhat", 3 = "Moderate", 4 = "Quite a bit", or 5 = "Extreme"). Total Symptom Score was calculated from this data by taking the sum of the intensity ratings from all 68 individual items using reverse scores for the three positive items from the list ("I Felt Good", "I Felt Alert", and "I Felt Wide Awake").
Sleep quality and quantify assessment during daylong exposure to indoor temperature limit. | At start of 8 hour daylong exposure.
  The Pittsburg Sleep Quality Index will be administered to provide an overview of the sleep quantity and quality of individuals over the previous month.

CONTACTS AND LOCATIONS:
Overall Officials: Glen Kenny, PhD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada